CLINICAL TRIAL: NCT06530576
Title: The Efficacy of Thalidomide for the Symptomatic Large Granular Lymphocytic Leukemia - a Prospective Phase Ⅱ Multicenter Clinical Trial From China
Brief Title: Thalidomide for the Symptomatic Large Granular Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024041
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: T-LGL Leukemia; NK-LGL Leukemia
Keywords: Large granular lymphocyte leukemia; Thalidomide; Overall response rate
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic | interventions — Thalidomide; Methotrexate

STUDY DESIGN:
Intervention Model Description: Thalidomide at a dose of 50-100 mg/QN
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalidomide (Experimental): All patients first receive thalidomide 100mg monotherapy.
  Interventions: Drug: Thalidomide and methotrexate

INTERVENTIONS:
Drug: Thalidomide and methotrexate — Thalidomide at a dose of 50-100 mg/QN, Methotrexate 10 mg/m2 orally once a week.

SUMMARY:
There is currently no standard first-line treatment for LGLL. The investigators used the TPM regimen (thalidomide + prednison + methotrexate ) to treat LGLL since 2020, enrolling a total of 54 patients and achieving an overall response rate (ORR) of 88.9% and a complete response (CR) rate of 75.9%. To further explore this hypothesis, the investigators designed this study to observe the efficacy of thalidomide monotherapy in patients with symptomatic LGLL. The investigators speculate that thalidomide plays a major role in the significant improvement of the TPM regimen compared to the MTX regimen.

Patients with LGLL are treated with thalidomide at 50 to 100 mg. If the desired response is not achieved at specific time points, methotrexate is added. Thalidomide monotherapy is administered for up to 3 courses, and the TM regimen can also be used for up to 3 courses. The overall response rate with thalidomide monotherapy serves as the primary study endpoint.

DETAILED DESCRIPTION:
The regimen is an oral treatment with a cycle of 4 months. All patients first receive monotherapy with thalidomide at a dose of 50-100 mg/QN. After 4 months, the efficacy is evaluated. If effective, the monotherapy continues for another 4 months. If complete remission (CR) is achieved, the treatment is consolidated for another 4 months before stopping, for a total of 3 courses. If CR is achieved at any point within the first year, the treatment is consolidated for one more course and then stopped. If partial remission (PR) is not achieved within the first cycle, or CR is not achieved within the second cycle, methotrexate 10 mg/m2 orally once a weekis a is dded for consolidation, with each cycle lasting 4 months. After a maximum of 3 cycles, treatment is stopped. Patients who do not achieve PR after 2 cycles of the TM regimen will be withdrawn from the study, with a maximum of 3 cycles allowed.

ELIGIBILITY:
Inclusion Criteria:

1. The patient fully understands the study, voluntarily participates, and signs the informed consent form (ICF);
2. The patient must meet the diagnostic criteria for LGLL;
3. The patient can be of any gender, aged 18 years or older;
4. The patient is either untreated or not properly treated previously, or has poor efficacy (not reaching PR) or relapsed after being treated with regimens not based on methotrexate/thalidomide;
5. The patient has indications for LGLL treatment, meeting at least one of the following criteria:

   1. ANC < 0.5 × 10^9/L, or neutropenia with recurrent infections
   2. HGB < 100 g/L or requiring red blood cell transfusions for maintenance
   3. PLT < 50 × 10^9/L
   4. Concurrent autoimmune disease requiring treatment
   5. Symptomatic splenomegaly
   6. Severe B symptoms (unexplained fever, temperature over 38°C; night sweats; weight loss of 10% or more within six months)
   7. Pulmonary hypertension;
6. ECOG score of 0-2;
7. The patient's expected survival period is 6 months or more.

Exclusion Criteria:

1. Unable to understand or follow the study procedures;
2. Diagnosed or treated for malignancies other than LGLL within the past five years;
3. Non-lymphoma-related liver or kidney function impairment: ALT > 3 times the upper limit of normal (ULN), AST > 3 times the ULN, total bilirubin (TBIL) > 2 times the ULN, serum creatinine clearance < 30 ml/min;
4. Other serious medical conditions that could affect the study (e.g., uncontrolled diabetes, gastric ulcer, other serious heart or lung diseases), with the judgment resting with the investigator;
5. Caprini thrombosis analysis score indicating high risk (Appendix 2);
6. Known history of HIV infection or active HBV infection, or any uncontrolled active systemic infection requiring intravenous antibiotics; Note: Active HBV infection is defined as: a. HBV DNA ≥ 2000 IU/ml; b. ALT ≥ 2 times the ULN; c. Exclusion of hepatitis due to the disease itself, drugs, or other causes. All three conditions must be met. If a patient initially has active HBV infection and turns into inactive HBV infection after anti-HBV treatment, they can be included in the study provided they receive adequate anti-HBV treatment.
7. Patients who have undergone major surgery (excluding lymph node biopsy) within the past 14 days or are expected to undergo major surgery during the treatment;
8. Pregnant or breastfeeding women, and women of childbearing age who are not using contraception;
9. Hypersensitivity to the drugs or their components used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 5 years
  complete remission rate+ partial remission rate

SECONDARY OUTCOMES:
The safety of thalidomide | up to 5 years
  Incidence of adverse events, serious adverse events and significant adverse event
Complete remession rate | up to 5 years
  Hematological PR was defined as an improvement in blood counts ANC > 0.5 × 109/L; HGB increased by >1 g/dL; PLT > 50 × 109/L
The rate of improvement in efficacy after TM combination | up to 5 years
  The effectiveness of the TM regimen is measured by subtracting the response rate of single-agent thalidomide
Progression-free survival | up to 5 years
  Progression-free survival
Overall survival | up to 5 years
  The time from the start of treatment to the patient's death from any cause
Duration of remission | up to 5 years
  the time from response to progression/death (P/D)

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No